CLINICAL TRIAL: NCT00913497
Title: Phase 4 Crossover Study Comparing the Effect of Insulin Glulisine to Insulin Aspart on Breakfast Post Prandial Blood Glucose Levels in Prepubertal Children With Type 1 Diabetes Mellitus on Multiple Daily Insulin Injection Therapy
Brief Title: The Effect of Insulin Glulisine Compared With Insulin Aspart on Breakfast Post Prandial Glucose Levels in Prepubertal Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Corewell Health West (Other)
Collaborators: Helen DeVos Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2009-089
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Results first posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 diabetes mellitus in children; insulin glulisine; insulin aspart; post prandial
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin glulisine; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- insulin glulisine (Active Comparator)
  Interventions: Drug: insulin glulisine
- insulin aspart (Active Comparator)
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: insulin glulisine — Insulin glulisine (Apidra®) Sanofi-Aventis; U100 (100 units/mL) 10 mL vials Prescribed dosage to be given subcutaneously at breakfast for a total of ten days
  Other Names: (Apidra®)
  Arms: insulin glulisine
Drug: insulin aspart — Insulin aspart (NovoLog®) Novo Nordisk; U100 (100 units/mL) 10 mL vials Prescribed dosage to be given subcutaneously at breakfast for a total of ten days.
  Other Names: (NovoLog®)
  Arms: insulin aspart

SUMMARY:
To determine whether insulin glulisine decreases the breakfast post prandial glycemic excursion in comparison to insulin aspart.

DETAILED DESCRIPTION:
This is a treatment, open label, crossover study comparing two and four hour breakfast post prandial blood glucose levels after receiving a dose of insulin glulisine or insulin aspart administered subcutaneously and consuming the breakfast meal from a prescribed menu containing 45, 60 or 75 grams of carbohydrate. Each subject will receive insulin glulisine for ten days and insulin aspart for ten days.

ELIGIBILITY:
Inclusion Criteria:

* current patient in the Helen DeVos Children's Hospital Diabetes Clinic;
* ages 4-11 years;
* prepubertal (Tanner Stage I);
* diagnosed with type 1 diabetes mellitus with positive islet cell antibodies or presenting at time of diagnosis with positive serum or urine ketones and requiring insulin since diagnosis;
* at least six months from date of diagnosis of type 1 diabetes mellitus;
* TSH within reference range and negative transglutaminase IgA antibodies within nine months of study start;
* HbA1C between 6.9 and 10% within 30 days of study start; parent or guardian able and willing to provide written informed consent prior to enrollment;
* at time of study start, current insulin regimen includes multiple daily injections with insulin glargine as the basal insulin and insulin aspart or insulin lispro as the pre-meal rapid acting insulin

Exclusion Criteria:

* pubertal (Tanner stage 2 or greater);
* concurrent Addison's disease, celiac disease or untreated hypothyroidism; - receiving oral, injectable or inhaled steroids or immunosuppressant medications;
* receiving stimulants for treatment of attention deficit disorder or attention deficit hyperactivity disorder;
* intercurrent illnesses such as a fever > 101 degrees F, infection, or gastroenteritis;
* use of any medication to treat diabetes other than those listed under in inclusion criteria;
* potential for lack of compliance or any other issue which, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2009-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayse P Cemeroglu, MD, Principal Investigator — Helen DeVos Childrens Hospital
Locations (1):
- Helen DeVos Childrens Hospital, Grand Rapids, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study is indicated to technically be a crossover study, however, participants were asked to take one medication on even days and the other on odd days. There was no washout period.
Groups:
- Insulin Glulisine and Insuline Asparte: insulin glulisine: Insulin glulisine (Apidra®) Sanofi-Aventis; U100 (100 units/mL) 10 mL vials. Insulin Asparte: (NovoLog®) Novo Nordisk; U100 (100 units/mL) 10 mL vials Prescribed dosage of insulin glulisine and aspart given subcutaneously at breakfast on alternate (10 days each for a total of 20 days)
Period: Overall Study
Arm/Group | Insulin Glulisine and Insuline Asparte
Started | 16
Completed | 13
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- All Participants: insulin glulisine: Insulin glulisine (Apidra®) Sanofi-Aventis; U100 (100 units/mL) 10 mL vials Prescribed dosage to be given subcutaneously at breakfast for a total of ten days insulin aspart: Insulin aspart (NovoLog®) Novo Nordisk; U100 (100 units/mL) 10 mL vials Prescribed dosage to be given subcutaneously at breakfast for a total of ten days.
Arm/Group | All Participants
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.8 (0.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 13
HbA1C [Mean (Standard Deviation); unit: percentage of total hemoglobin] | 7.7 (0.54)
BMI [Mean (Standard Deviation); unit: kg/m2] | 17.82 (2.47)

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Two Hour and Four Hour Post Prandial Blood Glucose Levels Following Administration of Insulin Glulisine Versus Insulin Aspart at the End of the Twenty Study Days
Description: Compare average blood glucose at 2 and 4 hours post prandial minus blood glucose at baseline (prior to eating)
Time Frame: measured daily at baseline, 2 and 4 hours post prandial for 20 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin Glulisine | Insulin Aspart
Number analyzed (Participants) | 13 | 13
mg/dL
  Baseline blood sugar (prior to eating) | 136.4 (15.7) | 133.4 (14.7)
  2 hour postprandial Blood Glucose excursion (2h measurement minus baseline) | 113.5 (65.2) | 98.6 (66.9)
  4 hour postprandial blood glucose excursion (4h measurement minus baseline) | 5.5 (36.5) | 4.4 (36.7)

2. Secondary Outcome: Occurrence of Hypoglycemia;
Time Frame: measured daily at 2 and 4 hours postprandial for 20 days
Population: analysis data is gathered from the published article, no further data is available
Measure: Number; unit: number of events
Arm/Group | Insulin Glulisine | Insulin Aspart
Number analyzed (Participants) | 13 | 13
number of events
  2 hour post prandial hypoglycemia | 8 | 9
  4 hour post prandial hypoglycemia | 19 | 26

ADVERSE EVENTS:
Time Frame: data gathered over 20 days of treatment. Participants alternated between study interventions for 10 days on each intervention.
Description: Adverse events were not specifically reported in the published work for this study. Patients in this study were members of both arms on alternating days.
Arm/Group | Insulin Glulisine | Insulin Aspart
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 8/13 | 9/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Glulisine (N=13) | Insulin Aspart (N=13)
hypoglycemia 2 hour postprandial (Endocrine disorders) | 4 (8) | 5 (9)
hypoglycemia 4 hours postprandial (Endocrine disorders) | 8 (19) | 9 (26)

LIMITATIONS AND CAVEATS:
This study was completed over 10 years ago, raw data is no longer available, the results reported in this entry are based on the published document for the trial that was published in 2013. This is the only information that is available for reporting. Per the published works, the target enrollment was met and data analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes